CLINICAL TRIAL: NCT03295526
Title: Study on Selective Pelvic Lymphadenectomy for IB-IIA Cervical Cancer
Brief Title: Selective Pelvic Lymphadenectomy for IB-IIA Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaohua Wu MD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STCSM2016-6-17-1.1
Record Dates: First submitted 2017-09-12; First posted 2017-09-28 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer, Lymph nodes debulking surgery
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): IB-IIA Cervical Cancer Patients with positive lymph node metastasis confirmed by intraoperative frozen pathological examination who will undergo radical hysterectomy and systematic pelvic lymphadenectomy
- Experimental group (Experimental): IB-IIA Cervical Cancer Patients with positive lymph node metastasis confirmed by intraoperative frozen pathological examination who will undergo radical hysterectomy and selective enlarged lymph node dissection.
  Interventions: Procedure: Lymph nodes debulking surgery.

INTERVENTIONS:
Procedure: Lymph nodes debulking surgery. — Radical hysterectomy and selective enlarged lymph node dissection
  Arms: Experimental group

SUMMARY:
Test name:

Study on selective pelvic lymphadenectomy for IB - IIA cervical cancer Researcher: Wu Xiaohua Research Center: Fudan University Shanghai Cancer Center The trial is expected to last for 3 years Test objectives： The primary goal：The overall therapeutic effect of patients with selective lymphadenectomy was not inferior to patients with systemic pelvic lymphadenectomy.

Secondary goal: Selective lymphadenectomy can reduce the incidence and severity of postoperative lower limb lymphedema.

The study was designed for prospective, randomized, controlled clinical trials. The number of subjects: 200 cases. Research groupings Selective pelvic lymphadenectomy group and The control group was treated with systematic pelvic lymph node dissection group.

Follow-up time: 3 years Sample size: 200 cases

End of the trial:

Primary end-poin:t three-year survival (overall survival, progression-free survival) Secondary end point: lower limb lymph node lymphedema

DETAILED DESCRIPTION:
Overall objective For cervical cancer patients with confirmed lymph node metastasis by intraoperative frozen pathology, the overall treatment effect of radical hysterectomy and selective enlarged lymph node dissection is not inferior to systematic pelvic lymphadenectomy and can reduce postoperative lower limb lymphedema incidence and severity.

1. The purpose of this study

1. to assess whether the progression free survival of patients with selective enlarged pelvic lymph node resection is better than patients with systematic pelvic lymph node dissection.
2. to evaluate differences of the incidence and severity of lymphedema between the two group patients using Lymphedema Staging standards (Stage 0-3) according to the"consensus document"of the International Society of Lymphology.

2. Preoperative evaluation LEEP, conization or biopsy Vagino-recto-abdominal examination + Vaginal / vaginal colposcopy examination History of Medical, surgical and childbearing Complications Physical condition Height and weight History of smoking Pregnancy test Chest X-ray or chest CT or general PET/CT Abdominal CT or general PET/CT Pelvic MRI/CT or general PET/CT

3.Protocol Patients with stage IB-IIa cervical cancer were randomly divided into two groups(Control group and Experimental group).Frozen pathological examination will be performed during the operation, and patients with positive lymph node metastasis will undergo radical hysterectomy and systematic pelvic lymphadenectomy or radical hysterectomy and selective enlarged lymph node dissection according to the patient's group.

4. Postoperative adjuvant therapy All patients with pelvic lymph node metastasis are required to receive DDP based concurrent chemoradiotherapy.

5.Efficacy evaluation Overall survival (OS): The period from randomization to death for any cause (for patients who have been loss to follow-up prior to death, the last follow-up time is calculated as the time of death).

Progression free survival (PFS): The duration from randomization to the earliest date of the date of tumor progression or the date of death for any cause. If the above standards are not met, the final evaluation date should be used for analysis.

Assessment of lymphedema in lower extremities: Lymphedema Staging standards (Stage 0-3) according to the"consensus document"of the International Society of Lymphology were used :

Stage 0 Subclinical with possible clinical evolution Stage I Edema regressing with treatments with positive pitting test Stage II Edema partially regressing with treatments with negative pitting test Stage III Elephantiasis with cutaneous complications and recurrent infections.

6. Follow up The patients were followed up every 3 months for the first year, every 4 months for the second year and every 6 months from the third year.

In addition to routine oncologic follow-up, the stage of patients̛ lower extremity lymphedema should also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. histology confirmed as cervical adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma.
2. histological grading of cervical cancer is 1, 2, 3 or not.
3. patients in the group must have no reproductive function requirements.
4. Patients must be ≥ 18 years of age.
5. preoperative: pelvic CT / MR or PET / CT suggest pelvic lymph node enlargement. Intraoperative: Patients with pelvic lymph node metastasis confirmed by freezing.
6. Signed informed consent.
7. Surgery should be completed within 4 weeks after the first diagnosis.
8. patients can receive treatment and follow-up.

Exclusion Criteria:

1. abdominal CT, PET / CT suggest that patients with para aortic lymph node metastasis.
2. other history of the tumor, but does not include: received appropriate treatment of non-melanoma skin cancer, has been cured of other solid tumors, has been cured or non Hodgkin's lymphoma and Hodgkin's lymphoma 5 years without recurrence.
3. Those who have received or will receive neoadjuvant chemotherapy.
4. patients with preoperative limb lymphedema or lower extremity venous and lymphatic reflux disorders.
5. pregnant women

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 3 year
  The period(months) from randomization to death for any cause (for patients who have been loss to follow-up prior to death, the last follow-up time is calculated as the time of death).

SECONDARY OUTCOMES:
Progression-Free-Survival (PFS) | 3 year
  The period(months) from randomization to the earliest date of the date of tumor progression or the date of death for any cause. If the above standards are not met, the final evaluation date should be used for analysis.
Lower extremities lymphedema | 3 year
  Lymphedema Staging standards (Stage 0-3) according to the"consensus document"of the International Society of Lymphology.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua WU, PhD & MD, Principal Investigator — Fudan university shanghai cancer center, Deparment of gynecologic oncology
Locations (1):
- Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No